CLINICAL TRIAL: NCT00577616
Title: Randomized Study Comparing Endovascular Repair Versus Conventional Repair for Ruptured Aorta-iliac Aneurysms
Brief Title: Ruptured Aorta-iliac Aneurysms: Endo vs. Surgery
Acronym: ECAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOM06055; K060216
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2013-07

CONDITIONS: Ruptured Aorta-iliac Aneurysms
Keywords: Endovascular repair; Ruptured aorta-iliac aneurysms; Mortality at 30 days
MeSH Terms: interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Endovascular repair
  Interventions: Procedure: Endovascular repair
- 2 (Other): conventional surgery repair
  Interventions: Procedure: Endovascular repair

INTERVENTIONS:
Procedure: Endovascular repair — Endovascular repair of the asymptomatic aneurysms of the abdominal aorta

SUMMARY:
The aim of this multicenter randomized trial is to compare the endovascular repair versus conventional repair for ruptured aorta-iliac aneurysms observed on CT scan in stable patients with suitable anatomy. The main awaited result is the significant reduction of the mortality of the conventional repair.

DETAILED DESCRIPTION:
The total death rate of ruptured aorta-iliac aneurysms is around 90%. A meta-analysis published by Bown et al. in 2002 in British Journal of Surgery finds on 171 studies compiled since 1955 an operational mortality post of the conventional surgery of 47%. This figure of post-operative mortality seems incompressible since many years in spite of the improvement of the techniques of anaesthesia and the surgery. The endovascular repair of the asymptomatic aneurysms of the abdominal aorta proved to be feasible and effective. In studies with limited and selected patients, the endovascular repair of ruptured aorta-iliac aneurysms seems to show a reduction in post-operative mortality in the average of 20%. However, the only comparative study (n=32) could not highlight of significant difference.This justifies a multicentric randomized study of which the goal is to compare the Endovascular repair and the Conventional repair in a cohort of a minimum of 160 patients carrying a Ruptured aorta-iliac Aneurysm(study name: ECAR) observed on CT-scan and being able to profit from the 2 techniques.The emergency does not allow the randomization by patient. The unit of randomization will be the week for each center, one week of endovascular treatment in alternation with one week of treatment by conventional repair and that in a synchronous way for the unit of all the centers of the study. The first week will be devoted to the conventional surgery and will be effective as of the opening of the first center. The principal objective is to compare mortality at 30 days in both groups. The secondary objectives are to compare in the 2 groups:• Morbidity (cardiac, pulmonary, renal, neurological, digestive) at 30 days.• Duration of stay in intensive care unit. The principal awaited results are a significant reduction in the mortality of the endovascular repair compared to the conventional surgery and a reduction in morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Ruptured aorta-iliac aneurysms diagnosed by CT
* scan with injection.
* Aneurysm developed on native infra-renal aorta or iliac.

  * Non infectious false aneurysms developed on prosthesis (Deleted by amendment n°1 at the request of AFSSAPS)
  * Ruptured aneurysm after endoprosthesis (Deleted by amendment n°1 at the request of AFSSAPS)
* Stable hemodynamic condition: systolic blood pressure on arrival higher than 80 mmHg in the absence of continuous vasopressive drugs administration.
* Anatomic criteria :length of aortic proximal neck >10 mm, diameter of aortic proximal neck < 32 mm, Absence of aortic neck angulation > 90° and patent iliac without important stenosis or tortuosity.
* Technical constraints (validation of experience form) : Trained operator (at least 15 endoprosthesis in asymptomatic patients), Endovascular materials at disposal

Exclusion Criteria:

* Unstable hemodynamic condition
* Anatomic criteria of non-inclusion
* Asymptomatic aneurysm
* Non-ruptured symptomatic aneurysm or aneurysm complicated with emboli.
* Mycotic aneurysm, infectious false aneurysms
* Post-traumatic aneurysm
* Supra-renal thoracic-abdominal aneurysm
* Impossibility to obtain a CT-scan with injection
* Patient non-affiliated to the social security and the protected people
* Pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-12; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Mortality at 30 days after the treatment(endovascular repair versus conventional repair) | 30 days after the treatment

SECONDARY OUTCOMES:
Compare at 30 days after the treatment the:- Cardiac , pulmonary, digestive , renal neurological morbidity, other…- Duration of stay in intensive care unit- Quantity of blood transfusions | 30 days after the treatment
Compare at 6 month after the treatment the:- Cardiac , pulmonary, digestive , renal neurological morbidity (amendment 6) | 6 month after treatment
Compare at one year after the treatment the:- Cardiac , pulmonary, digestive , renal neurological morbidity (amendment 6) | one year after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Desgranges, PUPH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHU Henri Mondor, Créteil, France

REFERENCES:
- [Background] Alsac JM, Desgranges P, Kobeiter H, Becquemin JP. Emergency endovascular repair for ruptured abdominal aortic aneurysms: feasibility and comparison of early results with conventional open repair. Eur J Vasc Endovasc Surg. 2005 Dec;30(6):632-9. doi: 10.1016/j.ejvs.2005.06.010. Epub 2005 Aug 1. PMID 16061405
- [Derived] Desgranges P, Kobeiter H, Katsahian S, Bouffi M, Gouny P, Favre JP, Alsac JM, Sobocinski J, Julia P, Alimi Y, Steinmetz E, Haulon S, Alric P, Canaud L, Castier Y, Jean-Baptiste E, Hassen-Khodja R, Lermusiaux P, Feugier P, Destrieux-Garnier L, Charles-Nelson A, Marzelle J, Majewski M, Bourmaud A, Becquemin JP; ECAR Investigators. Editor's Choice - ECAR (Endovasculaire ou Chirurgie dans les Anevrysmes aorto-iliaques Rompus): A French Randomized Controlled Trial of Endovascular Versus Open Surgical Repair of Ruptured Aorto-iliac Aneurysms. Eur J Vasc Endovasc Surg. 2015 Sep;50(3):303-10. doi: 10.1016/j.ejvs.2015.03.028. Epub 2015 May 20. PMID 26001320
- [Derived] Desgranges P, Kobeiter H, Castier Y, Senechal M, Majewski M, Krimi A. The Endovasculaire vs Chirurgie dans les Anevrysmes Rompus PROTOCOL trial update. J Vasc Surg. 2010 Jan;51(1):267-70. doi: 10.1016/j.jvs.2009.10.128. PMID 20117503